CLINICAL TRIAL: NCT03864185
Title: The Evaluation of Efficacy and Safety of Rituximab (Genetical Recombination) in Refractory Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Patients With Immunoglobulin G4 (IgG4) Autoantibodies in the Exploratory Clinical Trial
Brief Title: The Evaluation of Efficacy and Safety of Rituximab in Refractory CIDP Patients With IgG4 Autoantibodies
Acronym: RECIPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nagoya University (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government); Zenyaku Kogyo Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Masahiro Iijima, Designated Associate Professor, Nagoya University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAMCR-011; jRCT2041180037 (Registry Identifier: Japan Registry of Clinical Tials); UMIN000035753 (Registry Identifier: UMIN Clinical Trials Registry)
Record Dates: First submitted 2019-02-19; First posted 2019-03-06 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Keywords: IgG4 autoantibody; Neurofascin-155; Contactin-1; Rituximab
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rituximab group (IgG4 autoantibody positive) (Active Comparator)
  Interventions: Biological: Rituximab (genetical recombination)
- Placebo group (IgG4 autoantibody positive) (Placebo Comparator)
  Interventions: Other: Placebo
- Rituximab group (IgG4 autoantibody negative) (Active Comparator)
  Interventions: Biological: Rituximab (genetical recombination)

INTERVENTIONS:
Biological: Rituximab (genetical recombination) — Administer 375 mg/m2 of rituximab (genetical recombination) IV infusion once weekly for 4 doses.
  Arms: Rituximab group (IgG4 autoantibody negative); Rituximab group (IgG4 autoantibody positive)
Other: Placebo — Administer placebo IV infusion once weekly for 4 doses.
  Arms: Placebo group (IgG4 autoantibody positive)

SUMMARY:
To evaluate the efficacy and safety of rituximab (genetical recombination) intravenously administered to CIDP patients with positive or negative IgG4 autoantibody.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with definite CIDP diagnosed according to the modified diagnostic criteria of European Federation of Neurological Societies/Peripheral Nerve Society (EFNS/PNS) (2010) by the time of enrollment in the study
2. Patients meeting one of the following conditions:

   (i) Patients with positive serum IgG4 autoantibody (CNTN-1 or NF-155) confirmed by the time of enrollment in the study

   (ii) Patients with negative serum IgG4 autoantibody (CNTN-1 and NF-155) confirmed by the time of enrollment in the study
3. Patients with refractory CIDP not responding adequately to treatment with corticosteroid for 12 weeks, and intravenous immunoglobulin therapy (IVIg) for 8 weeks by the time of enrollment in the study, or those who are unable to administer or continue corticosteroid and IVIg
4. Patients with total adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Scale scores of 2 to 8 at both preliminary enrollment and enrollment, and with the total score at enrollment equal to or worse than that at preliminary enrollment
5. Patients aged 12 years or older at informed consent
6. Patients who give their voluntary written consent after having received adequate information on this study (legally acceptable representatives should also give consent for underage patients, and informed assent should be obtained from children aged 12 to 15)

Exclusion Criteria:

1. Patients with disease meeting one of the following exclusion criteria defined in the modified EFNS/PNS diagnostic criteria (2010).

   (i) Borrelia burgdorferi infection (Lyme disease), diphtheria, drug or toxin exposure probably to have caused the neuropathy Hereditary demyelinating neuropathy

   (ii) Prominent sphincter disturbance

   (iii) Diagnosis of multifocal motor neuropathy

   (iv) IgM monoclonal gammopathy with high titre antibodies to myelin-associated glycoprotein

   (v) Other causes for a demyelinating neuropathy including POEMS syndrome, osteosclerotic myeloma, diabetic and non-diabetic lumbosacral radiculoplexus neuropathy PNS lymphoma and amyloidosis may occasionally have demyelinating features
2. Patients who have started or have increased the dose of corticosteroid for CIDP within 12 weeks prior to the enrollment
3. Patients who have started or have increased the dose of IVIg within 8 weeks prior to the enrollment
4. Patients who have underwent plasmapheresis within 8 weeks prior to the enrollment or patients with refractory disease not responding adequately to 8 weeks of plasmapheresis (plasma exchange or double-filtration plasmapheresis)
5. Patients who have started or have increased the dose of an immunosuppressant (azathioprine, cyclophosphamide, cyclosporine, mycophenolate mofetil, interferon alpha, interferon beta, etanercept, methotrexate, mitoxantrone, alemtuzumab, cladribine, tacrolimus, fingolimod) within 12 weeks prior to the enrollment
6. Patients who have underwent hematopoietic stem cell transplant prior to the enrollment
7. Patients who have used rituximab (genetical recombination) prior to the enrollment
8. Patients who have participated in another clinical study within 3 months prior to the enrollment (enrollment is allowed for those participating in a clinical study in the range of Indications or Dosage and Administration in Japan) or patients who are participating in another study
9. Patients with poorly controlled diabetes (HbA1c of 7 % or higher)
10. Patients who have or are suspected to have active infection (infection requiring treatment with systemic antimicrobial, antifungal, or antiviral agents) at the time of the enrollment
11. Patients tested positive for HBs antigen, HBs antibody, HBc antibody, and/or HCV antibody (patients with positive HBs antibody or HBc antibody can be enrolled when a hepatitis B virus-DNA test is negative [below the limit of detection], and hepatitis B virus-DNA and aspartate/alanine transaminase levels are monitored at fixed intervals), or patients with positive HIV antibody or HTLV-1 antibody at the time of the enrollment
12. Patients with leukopenia (less than 2,000 /mm3), neutropenia (less than 1,000 /mm3), or lymphopenia (less than 500 /mm3) at the time of the enrollment
13. Patients with history of serious hypersensitivity or anaphylactic reaction to one of the ingredients in the investigational drug or murine protein-containing products
14. Patients with serious comorbidity (e.g., hepatic, renal, cardiac, lung, hematologic, or brain disease)
15. Female patients who are pregnant, lactating, or potentially pregnant, or patients who are not willing to use contraceptive measures during the study period
16. Patients who are judged to be unsuitable by the investigator or a sub-investigator

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-03-28 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-05-27 (Actual)

PRIMARY OUTCOMES:
Rate of patients with improvement in adjusted Inflammatory Neuropathy Cause and Treatment (INCAT) disability scale | Up to 52 weeks
  Primary analysis will compare scores of adjusted INCAT Disability Scale evaluated prior to treatment (at the time of enrollment) and scores at each timepoint after week 26 to calculate the proportion of patients who achieve an improvement of one and more from the baseline.
  The INCAT Disability Scale is an index to evaluate disorders in lower (gait) and upper (elevation of the upper arms and fine movement of the fingertips) extremities. The INCAT score is a 10-point scale and ranges from 0 (normal) to 10 (worst). For the "adjusted" INCAT score, a change in upper extremity score from 0 to 1 or 1 to 0 will not be considered meaningful in this evaluation.

SECONDARY OUTCOMES:
Change in grip strength (kPa) | Up to 52 weeks
  The differences of Grip strength (kPa) between prior to treatment and at each timepoint are summarized.
Change in Rasch-built Overall Disability Scale (R-ODS) score | Up to 52 weeks
  The differences of R-ODS score between prior to treatment and at each timepoint are summarized.
  R-ODS is consist of a 24-item questionnaire about daily living task with 3 response options: (0) "impossible to perform," (1) "performed with difficulty," and (2) "easily performed. The R-ODS score is a 48-point scale (range: 0-48), and is converted into a centile metric score with values ranging from 0 (most severe activity and social participation limitations) to 100 (no activity and social participation limitations).
Change in Medical Research Council (MRC) Sum Score | Up to 52 weeks
  The differences of MRC Sum Score between prior to treatment and at each timepoint are summarized.
  The MRC Sum Score is a scale to assess for 8 muscle groups (right and left side) as follow: Shoulder abduction, Elbow flexion, Wrist extension, Index finger abduction, Hip flexion, Knee extension, Foot dorsiflexion, Great toe dorsiflexion.The MRC Sum Score is a 80-point scale and ranges from 0 (paralysis) to 80 (normal strength).
Change in motor nerve distal latency | Up to 52 weeks
  The differences of distal latency between prior to treatment and at each timepoint are summarized.
Change in motor nerve proximal latency | Up to 52 weeks
  The differences of proximal latency between prior to treatment and at each timepoint are summarized.
Change in motor nerve compound muscle action potential (CMAP) | Up to 52 weeks
  The differences of CMAP between prior to treatment and at each timepoint are summarized.
Change in motor nerve conduction velocity | Up to 52 weeks
  The differences of motor nerve conduction velocity between prior to treatment and at each timepoint are summarized.
Cerebrospinal fluid protein level | Up to 52 weeks
  Cerebrospinal fluid protein level at each timepoint are summarized.
B cell counts (CD19 positive and CD20 positive cell counts) and T cell counts (CD3 positive, CD4 positive, and CD8 positive cell counts) | Up to 52 weeks
  B cell counts (CD19 positive and CD20 positive cell counts) and T cell counts (CD3 positive, CD4 positive, and CD8 positive cell counts) at each timepoint are summarized.
Expression of HACA | Up to 52 weeks
  The number of patients expressing HACA, and the proportion and its 95% confidence interval of these patients at each timepoint are summarized.
Serum rituximab (genetical recombination) level | Up to 52 weeks
  Serum rituximab (genetical recombination) level at each timepoint are summarized.
Maximum serum concentration (Cmax) of rituximab (genetical recombination) | Up to 52 weeks
  Cmax of rituximab (genetical recombination) is summarized.
Area under the curve (AUC) of blood concentration of rituximab (genetical recombination) | Up to 52 weeks
  AUC of blood concentration of rituximab (genetical recombination) is summarized.
Half-life (t1/2) of rituximab (genetical recombination) | Up to 52 weeks
  t1/2 of rituximab (genetical recombination) is summarized.
Clearance (CL) of rituximab (genetical recombination) | Up to 52 weeks
  CL of rituximab (genetical recombination) is summarized.
Mean residence time (MRT) of rituximab (genetical recombination) | Up to 52 weeks
  MRT of rituximab (genetical recombination) is summarized.
Volume of distribution (Vds) of rituximab (genetical recombination) level | Up to 52 weeks
  Vds of rituximab (genetical recombination) is summarized.
Serum antibody titers of IgG4 (CNTN-1 and NF-155) and these IgG subclass | Up to 52 weeks
  Serum titers (CNTN-1 and NF-155, and these IgG subclasses 1 to 4) at each timepoint are summarized.
Serum neurofilament | Up to 52 weeks
  Serum neurofilament level at each timepoint is summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Masahiro Iijima, Ph. D, Principal Investigator — Nagoya University Hospital
Locations (4):
- Japan (4):
  - Nagoya University Hospital, Nagoya, Aich
  - Chiba University Hospital, Chiba
  - Kyushu University Hospital, Fukuoka
  - Yamaguchi University Hospital, Ube

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shimizu S, Iijima M, Fukami Y, Tamura N, Nakatochi M, Ando M, Nishi R, Koike H, Kaida K, Koga M, Kanda T, Ogata H, Kira JI, Mori M, Kuwabara S, Katsuno M. Efficacy and Safety of Rituximab in Refractory CIDP With or Without IgG4 Autoantibodies (RECIPE): Protocol for a Double-Blind, Randomized, Placebo-Controlled Clinical Trial. JMIR Res Protoc. 2020 Apr 1;9(4):e17117. doi: 10.2196/17117. PMID 32234705